CLINICAL TRIAL: NCT06781190
Title: Promoting Mother-baby Bonding Through Sustainable Breastfeeding Practices: A Green Mom Approach
Brief Title: Promoting Mother-baby Bonding Through Sustainable Breastfeeding Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17.04.2024/43
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Attachment
Keywords: Sustainable Breastfeeding; Postpartum Attachment; Green Mom Initiative
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green motherhood education (Experimental): Pregnant women selected for the experimental group will receive 4 weeks of green motherhood training.
  The programme, which includes breastfeeding, bonding and carbon footprint training, is delivered 4 times by researchers.
  The training content has been prepared by the researchers by scanning the literature. The training will be delivered using posters.
  Interventions: Behavioral: Green motherhood education
- Standard of care (No Intervention): Women in the control group receive routine care at the same hospital's polyclinics.

INTERVENTIONS:
Behavioral: Green motherhood education — Pregnant women selected for the experimental group will receive 4 weeks of green motherhood training.
  Arms: Green motherhood education

SUMMARY:
This research aimed to identify sustainable breastfeeding practices and green mothers' initiatives to develop a strong mother-child bond.

DETAILED DESCRIPTION:
This research aimed to identify sustainable breastfeeding practices and green mothers' initiatives to develop a strong mother-child bond.

The sample size was calculated using G*Power 3.1. 9.7 software (Faul et al., 2007), the effect size was determined to be Cohen's d=0.9780770. Statistical power analysis was performed according to A Priori: Calculate required sample size (Means: Difference between two independent means (two groups)), 95% power (1-β) and α=0.05, and given these parameters it was concluded that a sample size of at least 58 participants was required for the study in question. In the event of data loss, a 20% increase in the sample size was expected as a result of statistical advice. Accordingly, it was planned to conduct the study with a total of n=70 people, n=35 in the intervention group and n=35 in the control group.

It was carried out with the participation of two groups. The green mother education group received 4 training sessions of 60 minutes each. The control group received routine hospital care but no other intervention during this period.

Data for the study were collected by the researcher using face-to-face interviews, a personal information form with demographic questions, and the measurement tools used in the study. The training was completed after 4 weeks. After the training, the measurement tools were used for the woman's postpartum period.

The participants were given an explanation of the green motherhood education and told how, for how long, and where the training would take place. The face-to-face green motherhood education programme was completed by the participants in a specific way for each session (nutrition, breastfeeding, environmental awareness and bonding). The training was delivered using a poster.

Green motherhood education was delivered in this way in 4 sessions. The measurement tools were given to the participants again on the 1st day, 1st month, 3rd month and 6th month after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 24 weeks gestation
* Must be between 18 and 35 years of age.
* Women must provide informed consent to participate in the study, indicating their willingness to participate in the educational intervention and assessments.
* Attend educational sessions
* Pregnant primiparous

Exclusion Criteria:

* Women with significant medical conditions that may affect breastfeeding or nutrition (e.g. serious mental illness, chronic disease) will be excluded.
* Multiple pregnancies
* Previous GREEN MOTHER training
* Substance abuse
* Women considered to be at high risk of non-compliance with the study protocol (e.g. those with unstable living conditions).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Famale
Enrollment: 100 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-01-18 (Actual)

PRIMARY OUTCOMES:
Sustainable and Healthy Eating Behaviors scale | Participants immediately after group assignment, 6 months after the birth
  The Sustainable and Healthy Eating Behaviours scale consists of 32 items and seven sub-dimensions. Quality labels (local and organic), seasonal food and avoiding food waste, animal health, reducing meat consumption, healthy and balanced diet, local food, low fat. Participants are asked to rate each item as 'never', 'very rarely', 'rarely', 'sometimes', 'often', 'very often' or 'always'. Never' is worth 1 point and 'always' is worth 7 points. Factor scores are calculated by taking the average of the scores given to the items in that factor (between 1 and 7 points). Cronbach's alpha was found to be 0.912.
  The lowest possible score is 32 and the highest is 224. This reflects high sustainability.
Carbon Footprint Awareness Scale | Participants immediately after group assignment, 6 months after the birth
  The scale comprises 19 items measured on a 5-point Likert-type scale, focusing on five key areas: transportation, which includes 3 items; fuel consumption, also with 3 items; electricity use, featuring 5 items; food consumption, containing 5 items; and waste management, which has 3 items. The scale demonstrates a strong factor structure, with a Cronbach's alpha of 0.86, indicating high reliability, and it explains 56.09% of the variance in the data. The lowest score is 19 and the highest is 95. High scores indicate sustainability.
Depression Anxiety and Stress scales-21 | Participants immediately after group assignment, 1st day after delivery, 3rd month after delivery, 6th month after delivery
  This 21-item scale consists of three dimensions, namely anxiety, depression, and stress. Items are measured on a 4-point Likert-type scale ranging from 0 (Never) to 3 (Always). A higher sum score indicates more severe symptoms of depression, anxiety, and stress.
Multidimensional Scale of Perceived Social Support | Participants were assigned to the group immediately after birth, 1 day after birth, 3 months after birth and 6 months after birth.
  Multidimensional Scale of Perceived Social Support is a psychometric tool designed by Zimet et al. 18 and adapted to Turkish by Eker et al. 19 to measure individuals' perceived social support from three sources: "family, friends, and a significant other." This scale comprises 12 items, rated on a 5-point Likert-type scale from strongly disagree to strongly agree. The internal consistency coefficients reported for the scale are within the range of 0.80 to 0.85, with a Cronbach's alpha coefficient of 0.92.
Scale Breast-feeding Self-efficacy Scale | 1st day after birth, 3rd month after birth, 6th month after birth
  Breastfeeding Self-Efficacy Scale: This is a 33-item scale developed by Dennis (1999). It consists of two sub-dimensions to determine mothers' breastfeeding skills, beliefs and behaviours regarding breastfeeding. The validity and reliability study of the Turkish form of the scale was conducted by Ekşioğlu and Çeber (2011). Breastfeeding self-efficacy was assessed using a five-point Likert scale: (1) I never trust myself, (2) I do not trust myself very much, (3) I trust myself sometimes, (4) I trust myself often, (5) I always trust myself. As the total score on the scale increases, so does breastfeeding self-efficacy. The lowest score is 33 and the highest is 165.
Postpartum Attachment Scale | 1st day after birth, 3rd month after birth, 6th month after birth
  The Postpartum Attachment Scale is a mother-filled assessment tool that utilizes a six-point Likert scale defined as "always," "very often," "often," "sometimes," "rarely," and "never." This scale consists of 25 items, with some items rated inversely, and scores range from 0 to 5. It is organized into four sub-dimensions: "attachment disorder" with 12 items, "rejection and irritability" with 7 items, "tension about care" with 4 items, and "risk of abuse" with 2 items. The overall cut-off point for the scale is set at 26 points, with a score of 27 or above indicating a postpartum attachment problem. In the original study, the total score had a Cronbach's alpha of 0.75, while the subscales showed varying reliability: 0.62 for attachment disorder, 0.53 for rejection and irritability, 0.40 for anxiety in babysitting, and 0.11 for risk of abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kaya, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Esra Keles, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)